CLINICAL TRIAL: NCT00437671
Title: Pharmacokinetics Of Active And Passive Tetanus Immunization Given Concurrently In Subjects With No Known Primary Immunization History Or In Subjects With Tetanus Antibody Levels Below Protective Levels
Brief Title: Tetanus Immunization in Subjects With No Immunization History or With Tetanus Antibody Levels Below Protective Levels
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study terminated for cGCP non-compliance. Analyses could not be performed.
Sponsor: Grifols Therapeutics LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 060002
Record Dates: First submitted 2007-02-20; First posted 2007-02-21 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Tetanus
Keywords: trismus; lockjaw
MeSH Terms: conditions — Tetanus; Trismus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Entered study (Experimental)
  Interventions: Drug: Tetanus Immune Globulin (Human); Biological: Diphtheria-Tetanus Toxoids Adsorbed

INTERVENTIONS:
Drug: Tetanus Immune Globulin (Human) — Based on package insert recommendation and recommendations of WHO
  Other Names: HyperTET S/D; BayTet; BAY 19-8515; TAL-05-00013; NDC 13533-634-02
Biological: Diphtheria-Tetanus Toxoids Adsorbed — Based on package insert recommendations and recommendations of WHO

SUMMARY:
The goal of this study is to re-evaluate the tetanus antibody pharmacokinetic profile when Tetanus Immune Globulin (Human)(TIG) and Tetanus vaccine (Tetanus toxoid; TT) are given concurrently with strict control on the anatomical location and timing of administration of TIG and TT. Pharmacokinetic profile of antibody titer including the duration of adequate titer protection provided by TIG and TT given in combination will be assessed using a standardized administration regimen and standardized antibody assay procedure. This study may provide evidence for the recommendations of the World Health Organisation (WHO) whereby dual coverage with both a vaccine and tetanus hyperimmune would ideally provide the best coverage for anyone with the potential of developing tetanus.

DETAILED DESCRIPTION:
This is a prospective, open-label, single-center trial including a single group of subjects with no known primary immunization history with TT or >10 years have passed since the last dose of tetanus containing vaccine was received. The study will enroll six subjects who would receive both dT and TIG concurrently on Day 1.

All dosed subjects will be followed for 40 days during which Day 1, 2, 3, 4, 5, 7, 14, 21, 30 and 40 time levels of tetanus antibodies will be measured in order to determine the serum level vs. time curve, Cmax, Tmax, and duration of protective antibody levels.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 90 years.
* Signed a written informed consent prior to initiation of any study-related procedures.
* No known primary immunization history with TT/dT or >10 years have passed since the last dose of tetanus containing vaccine was received. Subjects with unknown or uncertain previous vaccination histories are considered to have no previous tetanus and toxoid doses. Subjects who have had military service since 1941 will be considered to have had 1 dose of tetanus vaccine.
* Subjects must have documented tetanus antibody levels that are non-protective levels (< 0.15 IU/ml).
* Subjects must be free of any presenting wound or wound infection

Exclusion Criteria:

* History or suspicion of significant allergic reaction to intravenous immune globulin, and or blood products
* A history of selective IgA deficiency (serum level <5.0 mg/dL) and known antibodies to IgA
* Congestive heart failure (New York Association stage greater than Class II)
* Conditions whose symptoms and effects could alter protein catabolism and/or IgG utilization (e.g. protein-losing enteropathies, nephrotic syndrome)
* Women of child bearing potential who do not practice adequate contraception (i.e. chemical or mechanical methods) and pregnant or lactating females
* Subjects who have severe thrombocytopenia or any coagulation disorder that would contraindicate intramuscular injections
* TIG therapy within the previous six months
* Investigational drug therapy within the previous three months
* History of Thromboembolism

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2007-03; Primary Completion 2007-09 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Antibody titer serum level at each time point | 40 days
Cmax | 40 days
Tmax | 40 days

CONTACTS AND LOCATIONS:
Overall Officials: Kumar Alagappan, MD, Principal Investigator — Long Island Jewish Medical Center
Locations (1):
- Long Island Jewish Medical Center, New Hyde Park, New York, United States

REFERENCES:
- Available data/document: FDA approved labeling information — http://www.talecris-pi.info/inserts/hypertet.pdf